CLINICAL TRIAL: NCT03515681
Title: Retail Outlet Health Kiosk Hypertension Trial
Acronym: ROKHyT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Higi (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven J. Shea, Professor of Medicine and Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAR3975; 5R34HL137659 (NIH)
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
Keywords: Text messaging
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects randomized to intervention will receive text messages to promote seeking care and improving compliance with blood pressure treatment.
  Interventions: Behavioral: Text messages
- Control (No Intervention): Subjects randomized to the control arm will receive the messages regarding their kiosk blood pressure levels currently provided by higi to kiosk users. These messages are provided at the kiosk at the time of the blood pressure measurement (no text messages).

INTERVENTIONS:
Behavioral: Text messages — Subjects randomized to intervention will receive text messages to promote seeking care and improving compliance with blood pressure treatment.
  Arms: Intervention

SUMMARY:
The investigators propose to conduct pilot studies to support an application to conduct a fully powered randomized trial of a text messaging intervention to increase the rate of blood pressure control, defined as <140/90 mmHg, among hypertensive individuals using health kiosk blood pressure devices. These pilot studies will include testing of the intervention, recruitment, enrollment, and data collection procedures, and of the web-based interactions between the data coordinating center and higi Sh llc (Chicago, IL), which is the company that installs and maintains the health care kiosks and associated software infrastructure. Completion of these pilot studies will provide preliminary data to support an application for a full scale randomized controlled study. Potential for adaption is high because of alignment of retail outlets, kiosk providers, and consumers for health, wellness, and self-care.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains the leading cause of death in the U.S. as well as the leading cause of health care cost. Hypertension is the leading remediable risk factor for CVD in the U.S. and globally, with prevalence of 29% in U.S. adults. Recent data from NHANES indicate that blood pressure (BP) is not controlled, defined as <140/90 mmHg, in 48% of individuals in the U.S. with hypertension. Strategies to improve hypertension control have focused on the physician-patient interaction at the office visit, system factors in the health care provider system, and extension beyond the traditionally defined health care system. All have had some success but are limited by not reaching individuals outside the clinical encounter or by challenges of scale, scope, and standardization of blood pressure measurement outside the clinical setting. Retail outlet BP devices have the potential to address these limitations by providing free BP measurements to individuals outside the clinical setting and at all times the retail outlet is open. These automated devices are standardized and linked to software with the ability to collect data and provide information to individuals using these devices, thereby providing a platform for an intervention strategy. Higi is a privately owned company that provides health kiosks in retail outlets. Higi presently has 10,800 kiosks in the U.S. with 4,125 in Rite Aid pharmacies. More than 44 million BP measurements per year are obtained at higi kiosks. In the one-year period 7/1/15 to 6/30/16, approximately 727,000 individuals using higi kiosks recorded >3 systolic BP measurements >140/90 mmHg. The investigators propose to target this group using interactive text messaging to activate individuals to take actions to improve BP control. The primary endpoint will be BP control defined as <140/90 mmHg at 12 months post randomization.

ELIGIBILITY:
Inclusion Criteria:

* >3 systolic blood pressure measurements >140/90 mmHg (two in the previous 12 months + one at baseline)
* Age 18-85 years
* Weight <300 pounds
* Has a cell phone
* Can provide consent
* Speaks English or Spanish

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shea, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shea S, Thompson JLP, Schwartz JE, Chen Y, de Ferrante M, Vanderbeek AM, Buchsbaum R, Vargas C, Siddiqui KM, Moran AE, Stockwell M. The Retail Outlet Health Kiosk Hypertension Trial (ROKHYT): Pilot Results. Am J Hypertens. 2022 Jan 5;35(1):103-110. doi: 10.1093/ajh/hpab129. PMID 34382648
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 70 | 70
Randomized | 70 | 70
Completed at 6 Months | 61 | 62
Completed (Completed at 12 months) | 37 | 25
Not Completed | 33 | 45

BASELINE CHARACTERISTICS:
Population: Only the randomized participants are counted in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (12.2) | 51.4 (11.2) | 52.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 36 | 37 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 61 | 58 | 119
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 51 | 48 | 99
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 4 | 9 | 13
Mean systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 146.7 (20.6) | 144.4 (17.0) | 145.5 (18.9)
Mean diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 92.2 (12.2) | 91.3 (12.7) | 91.8 (12.4)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants With Blood Pressure Control at 12 Months
Description: Blood pressure (BP) control is defined as having BP <140/90 mmHg.
Time Frame: 12 months after randomization
Population: Only includes individuals who completed the study at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 25
Participants | 13 | 7

2. Secondary Outcome: Total Number of Participants With Blood Pressure Control at 6 Months
Description: Blood pressure (BP) control is defined as having BP <140/90 mmHg.
Time Frame: 6 months
Population: Only includes participants who completed the study at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 61 | 62
Participants | 22 | 19

3. Secondary Outcome: Total Number of Participants With Blood Pressure Control at 3 Months
Description: Blood pressure (BP) control is defined as having BP <140/90 mmHg.
Time Frame: 3 months
Population: Only includes participants who completed the study at 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 67 | 64
Participants | 24 | 20

4. Secondary Outcome: Mean Systolic Pressure at 12 Months
Description: Mean systolic blood pressure measurement at 12 months from randomization.
Time Frame: 12 months
Population: Only includes participants who completed the study at 12 months.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 25
mm Hg | 141.2 (17.91) | 147.0 (19.65)

5. Other Pre Specified Outcome: Study Participation Rate
Description: Proportion of those invited to participate who consent and are randomized.
Time Frame: 2 weeks
Population: Includes all consented individuals.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 78 | 72
Participants | 70 | 70

6. Other Pre Specified Outcome: Study Completion Rate
Description: Proportion of those randomized who completed follow up at month 6.
Time Frame: 6 months
Population: Only includes randomize participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 70 | 70
Participants | 61 | 62

7. Secondary Outcome: Mean Diastolic Pressure at 12 Months
Description: Mean diastolic blood pressure measurement at 12 months from randomization.
Time Frame: 12 months
Population: Only includes individuals who completed the study at 12 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 25
mm Hg | 88.0 (11.90) | 88.8 (12.73)

ADVERSE EVENTS:
Time Frame: Up to 12 months from Baseline
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT03515681/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT03515681/SAP_001.pdf